CLINICAL TRIAL: NCT01287117
Title: A Phase III, Multicenter, Randomized, Double-blind, Placebo-controlled, Dose-ranging Study to Evaluate the Efficacy and Safety of Xolair® (Omalizumab) in Patients With Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite Antihistamine Treatment (H1)
Brief Title: A Study of the Efficacy and Safety of Omalizumab (Xolair) in Patients With Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) Who Remain Symptomatic Despite Antihistamine (H1) Treatment
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Q4881g; GA00887
Record Dates: First submitted 2011-01-27; First posted 2011-02-01 (Estimated); Results first posted 2013-10-18 (Estimated); Last update posted 2013-11-27 (Estimated); Status verified 2013-11

CONDITIONS: Chronic Idiopathic Urticaria
MeSH Terms: conditions — Chronic Urticaria | interventions — Omalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (4):
- Placebo (Placebo Comparator): Participants received placebo subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Placebo
- Omalizumab 75 mg (Experimental): Participants received omalizumab 75 mg subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Omalizumab
- Omalizumab 150 mg (Experimental): Participants received omalizumab 150 mg subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Omalizumab
- Omalizumab 300 mg (Experimental): Participants received omalizumab 300 mg subcutaneously every 4 weeks during the 24 week treatment period.
  Interventions: Drug: Omalizumab

INTERVENTIONS:
Drug: Omalizumab — Omalizumab was supplied as a lyophilized, sterile powder in a single-use vial.
  Other Names: Xolair
  Arms: Omalizumab 150 mg; Omalizumab 300 mg; Omalizumab 75 mg
Drug: Placebo — Placebo was supplied as a lyophilized, sterile powder in a single-use vial without study drug.
  Arms: Placebo

SUMMARY:
The study is a global Phase III, multicenter, randomized, double-blind, placebo-controlled, parallel-group study to evaluate the efficacy and safety of omalizumab administered subcutaneously as an add-on therapy for the treatment of adolescent and adult patients aged 12-75 who have been diagnosed with refractory CIU and who remain symptomatic despite standard-dose H1 antihistamine treatment.

DETAILED DESCRIPTION:
Type I Error Rate Control Plan

Primary Outcome Measure

In order to maintain an overall type I error rate of 0.05 (2-sided) across the 3 omalizumab dose levels, the testing of the primary Outcome Measure was conducted in the following hierarchical order. A p-value < 0.05 is only considered statistically significant if statistical significance was claimed at the previous stage.

* Stage 1: Omalizumab 300-mg group vs. placebo
* Stage 2: Omalizumab 150-mg group vs. placebo
* Stage 3: Omalizumab 75-mg group vs. placebo

Secondary Outcome Measures

A hierarchical analysis of the following secondary Outcome Measures was performed for each dose found to be significant in the primary Outcome Measure. A p-value < 0.05 is only considered statistically significant if statistical significance was claimed at the previous stage.

* Stage 1: Change from baseline to Week 12 in the urticaria activity score over 7 days (UAS7)
* Stage 2: Change from Baseline to Week 12 in the weekly number of hives score
* Stage 3: Time to minimally important difference (MID) response in the weekly itch severity score by Week 12
* Stage 4: Percentage of participants with a UAS7 score ≤ 6 at Week 12
* Stage 5: Percentage of weekly itch severity score MID responders at Week 12
* Stage 6: Change from Baseline to Week 12 in the weekly size of the largest hive score
* Stage 7: Change from Baseline in the overall dermatology life quality index (DLQI) score at Week 12
* Stage 8: Change from Baseline in the overall dermatology life quality index (DLQI) score at Week 12
* Stage 9: Percentage of complete responders (UAS7 = 0) at Week 12

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Chronic Idiopathic Urticaria (CIU)/Chronic Spontaneous Urticaria (CSU) refractory to H1 antihistamines at the time of randomization.

Exclusion Criteria:

* Treatment with an investigational agent within 30 days prior to screening.
* Weight < 20 kg (44 lbs).
* Clearly defined underlying etiology for chronic urticarias other than CIU.
* Evidence of parasitic infection.
* Atopic dermatitis, bullous pemphigoid, dermatitis herpetiformis, senile pruritus, or other skin disease associated with itch.
* Previous treatment with omalizumab within a year prior to screening.
* Routine doses of the following medications within 30 days prior to screening: Systemic or cutaneous (topical) corticosteroids (prescription or over the counter), hydroxychloroquine, methotrexate, cyclosporine, or cyclophosphamide.
* Intravenous (IV) immunoglobulin G (IVIG), or plasmapheresis within 30 days prior to screening.
* Regular (daily/every other day) doxepin (oral) use within 6 weeks prior to screening.
* Any H2 antihistamine use within 7 days prior to screening.
* Any leukotriene receptor antagonist (LTRA) (montelukast or zafirlukast) within 7 days prior to screening.
* Any H1 antihistamines at greater than approved doses within 3 days prior to screening.
* Patients with current malignancy, history of malignancy, or currently under work-up for suspected malignancy except non-melanoma skin cancer that has been treated or excised and is considered resolved.
* Hypersensitivity to omalizumab or any component of the formulation.
* History of anaphylactic shock.
* Presence of clinically significant cardiovascular, neurological, psychiatric, metabolic, or other pathological conditions that could interfere with the interpretation of the study results and or compromise the safety of the patients.
* Evidence of current drug or alcohol abuse.
* Nursing women or women of childbearing potential, unless they meet the following definition of post-menopausal: 12 months of natural amenorrhea or 6 months of spontaneous amenorrhea with serum follicle-stimulating hormone (FSH) levels > 40 mIU/mL or 6 weeks post surgical bilateral oophorectomy (with or without hysterectomy) or hysterectomy or are using one or more of the following acceptable methods of contraception: surgical sterilization, hormonal contraception, and double-barrier methods.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 319 (Actual)
Dates: Start 2011-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (63):
- United States (40):
  - Birmingham, Alabama
  - Huntington Beach, California
  - Long Beach, California
  - Los Angeles, California
  - Palmdale, California
  - Sacramento, California
  - San Jose, California
  - Studio City, California
  - Centennial, Colorado
  - Washington D.C., District of Columbia
  - Coral Gables, Florida
  - Sarasota, Florida
  - Tallahassee, Florida
  - Columbus, Georgia
  - Springfield, Illinois
  - Indianapolis, Indiana
  - Baltimore, Massachusetts
  - Boston, Massachusetts
  - Burlington, Massachusetts
  - St Louis, Missouri
  - Edison, New Jersey
  - Skillman, New Jersey
  - Staten Island, New York
  - The Bronx, New York
  - Durham, North Carolina
  - Columbus, Ohio
  - Toledo, Ohio
  - Tulsa, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Upland, Pennsylvania
  - Charleston, South Carolina
  - Fort Worth, Texas
  - Houston, Texas
  - Waco, Texas
  - Salt Lake City, Utah
  - Sandy City, Utah
  - Springfield, Virginia
  - La Crosse, Wisconsin
  - Madison, Wisconsin
- Denmark (2):
  - Copenhagen
  - Odense
- France (3):
  - Bordeaux
  - Marseille
  - Reims
- Germany (6):
  - Berlin
  - Dresden
  - Freiburg im Breisgau
  - Heidelberg
  - München
  - Münster
- Italy (3):
  - Perugia
  - Roma
  - Terni
- Poland (4):
  - Krakow
  - Lodz
  - Lublin
  - Wroclaw
- Spain (2):
  - Barcelona
  - Pamplona
- Turkey (Türkiye) (3):
  - Ankara
  - Bursa
  - Istanbul

REFERENCES:
- [Derived] Casale TB, Trzaskoma B, Holden M, Bernstein JA, Maurer M. Does angioedema in patients with chronic spontaneous urticaria impact response to omalizumab? World Allergy Organ J. 2024 Aug 5;17(8):100943. doi: 10.1016/j.waojou.2024.100943. eCollection 2024 Aug. PMID 39193419
- [Derived] Ferrer M, Gimenez-Arnau A, Saldana D, Janssens N, Balp MM, Khalil S, Risson V. Predicting Chronic Spontaneous Urticaria Symptom Return After Omalizumab Treatment Discontinuation: Exploratory Analysis. J Allergy Clin Immunol Pract. 2018 Jul-Aug;6(4):1191-1197.e5. doi: 10.1016/j.jaip.2018.04.003. Epub 2018 Apr 12. PMID 29655772
- [Derived] Goldstein S, Gabriel S, Kianifard F, Ortiz B, Skoner DP. Clinical features of adolescents with chronic idiopathic or spontaneous urticaria: Review of omalizumab clinical trials. Ann Allergy Asthma Immunol. 2017 Apr;118(4):500-504. doi: 10.1016/j.anai.2017.02.003. PMID 28390587
- [Derived] Saini SS, Omachi TA, Trzaskoma B, Hulter HN, Rosen K, Sterba PM, Courneya JP, Lackey A, Chen H. Effect of Omalizumab on Blood Basophil Counts in Patients with Chronic Idiopathic/Spontaneous Urticaria. J Invest Dermatol. 2017 Apr;137(4):958-961. doi: 10.1016/j.jid.2016.11.025. Epub 2016 Dec 6. No abstract available. PMID 27939380
- [Derived] Gimenez-Arnau AM, Spector S, Antonova E, Trzaskoma B, Rosen K, Omachi TA, Stull D, Balp MM, Murphy T. Improvement of sleep in patients with chronic idiopathic/spontaneous urticaria treated with omalizumab: results of three randomized, double-blind, placebo-controlled studies. Clin Transl Allergy. 2016 Aug 18;6:32. doi: 10.1186/s13601-016-0120-0. eCollection 2016. PMID 27540466
- [Derived] Zazzali JL, Kaplan A, Maurer M, Raimundo K, Trzaskoma B, Solari PG, Antonova E, Mendelson M, Rosen KE. Angioedema in the omalizumab chronic idiopathic/spontaneous urticaria pivotal studies. Ann Allergy Asthma Immunol. 2016 Oct;117(4):370-377.e1. doi: 10.1016/j.anai.2016.06.024. Epub 2016 Jul 14. PMID 27424128
- [Derived] Casale TB, Bernstein JA, Maurer M, Saini SS, Trzaskoma B, Chen H, Grattan CE, Gimenez-Arnau A, Kaplan AP, Rosen K. Similar Efficacy with Omalizumab in Chronic Idiopathic/Spontaneous Urticaria Despite Different Background Therapy. J Allergy Clin Immunol Pract. 2015 Sep-Oct;3(5):743-50.e1. doi: 10.1016/j.jaip.2015.04.015. Epub 2015 Jun 6. PMID 26054553
- [Derived] Saini SS, Bindslev-Jensen C, Maurer M, Grob JJ, Bulbul Baskan E, Bradley MS, Canvin J, Rahmaoui A, Georgiou P, Alpan O, Spector S, Rosen K. Efficacy and safety of omalizumab in patients with chronic idiopathic/spontaneous urticaria who remain symptomatic on H1 antihistamines: a randomized, placebo-controlled study. J Invest Dermatol. 2015 Jan;135(1):67-75. doi: 10.1038/jid.2014.306. Epub 2014 Jul 21. PMID 25046337

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomized population: All randomized participants regardless of whether they received any study drug.
Period: Overall Study
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Started | 80 | 78 | 80 | 81
Received Treatment | 80 | 77 | 80 | 81
Completed | 65 | 64 | 64 | 69
Not Completed | 15 | 14 | 16 | 12
Not completed — Adverse Event | 2 | 1 | 1 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 1 | 1
Not completed — Patient/Legal Guardian's Decision | 2 | 6 | 8 | 5
Not completed — Disease Progression | 10 | 5 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Modified intent-to-treat (mITT) population: All participants randomized in the study who received at least 1 dose of study drug. 1 participant (randomized to omalizumab 75 mg) did not receive study drug and was not included in the mITT population.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg | Total
Number analyzed (Participants) | 80 | 77 | 80 | 81 | 318
Age Continuous [Mean (Standard Deviation); unit: years] | 40.4 (15.6) | 40.7 (15.2) | 41.1 (14.0) | 42.4 (13.2) | 41.2 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 64 | 60 | 231
  Male | 28 | 22 | 16 | 21 | 87

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Weekly Itch Severity Score
Description: The weekly itch severity score is the sum of the daily itch severity scores over 7 days and ranges from 0 to 21. The daily itch severity score is the average of the morning and evening scores on a scale of 0 (none) to 3 (severe). The Baseline weekly itch severity score is the sum of the daily itch severity scores over the 7 days prior to the first treatment. A higher itch severity score indicates more severe itching. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Units on a scale | -3.63 (5.22) | -6.46 (6.14) | -6.66 (6.28) | -9.40 (5.73)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0010, ANCOVA — A multiplicity type I error control plan was employed to adjust for the comparison of multiple omalizumab groups to the placebo group in order to maintain an overall type I error rate of 0.05 (2-sided); Covariates included in the analysis were baseline weekly itch severity score (< 13 vs ≥ 13) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -2.96, 95% CI 2-sided [-4.71 to -1.21]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0012, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -2.95, 95% CI 2-sided [-4.72 to -1.18]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = -5.80, 95% CI 2-sided [-7.49 to -4.10]

2. Secondary Outcome: Change From Baseline to Week 12 in the Urticaria Activity Score Over 7 Days (UAS7)
Description: The UAS7 is the sum of the daily urticarial activity scores over 7 days and ranges from 0 to 42. The daily urticarial activity score is the average of the morning and evening urticarial activity scores and ranges from 0 to 6. The urticarial activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticarial activity scores over the 7 days prior to the first treatment. A higher urticarial activity score indicates more urticaria activity. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Units on a scale | -8.01 (11.47) | -13.82 (13.26) | -14.44 (12.95) | -20.75 (12.17)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0035, ANCOVA — A pre-specified hierarchical order of testing was employed to adjust for the comparison of multiple omalizumab groups to the placebo group in order to maintain an overall type I error rate of 0.05 (2-sided) within each dose; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -5.75, 95% CI 2-sided [-9.59 to -1.92]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0008, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -6.54, 95% CI 2-sided [-10.33 to -2.75]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -12.80, 95% CI 2-sided [-16.44 to -9.16]

3. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Number of Hives Score
Description: The weekly hives score is the sum of the daily hives scores over 7 days and ranges from 0 to 21. The number of hives is measured twice daily (morning and evening) on a scale of 0 (none) to 3 (> 12 hives per 12 hours). The daily hives score is the average of the morning and evening scores. The Baseline score is the sum of the daily hives scores over the 7 days prior to the first treatment. A higher score indicates more hives. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Units on a scale | -4.37 (6.60) | -7.36 (7.52) | -7.78 (7.08) | -11.35 (7.25)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0149, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline weekly number of hives score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -2.75, 95% CI 2-sided [-4.95 to -0.54]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0017, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]; Least squares mean difference = -3.44, 95% CI 2-sided [-5.57 to -1.32]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 3, analysis 1]; Least squares mean difference = -6.93, 95% CI 2-sided [-9.10 to -4.76]

4. Secondary Outcome: Time to Minimally Important Difference (MID) Response in the Weekly Itch Severity Score by Week 12
Description: The time to the MID response is the number of weeks from the start of treatment (Baseline) until the time point at which the first MID response occurs. The MID response is defined as a reduction ≥ 5 points from Baseline in the weekly itch severity score.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 57 | 57 | 66 | 76
Weeks | 4.0 [2.0 to 6.0] | 3.0 [2.0 to 5.0] | 2.0 [2.0 to 3.0] | 1.0 [1.0 to 2.0]
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 75 mg groups; Test type: Superiority or Other; p = 0.0879, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [0.95 to 2.03]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0301, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 1.49, 95% CI 2-sided [1.04 to 2.14]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cox proportional hazards model — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]; Hazard Ratio (HR) = 2.34, 95% CI 2-sided [1.63 to 3.36]

5. Secondary Outcome: Percentage of Participants With a UAS7 Score ≤ 6 at Week 12
Description: The UAS7 is the sum of the daily urticarial activity scores over 7 days and ranges from 0 to 42. The daily urticarial activity score is the average of the morning and evening urticarial activity scores and ranges from 0 to 6. The urticarial activity score is the sum of ratings on a scale of 0 to 3 (0=none to 3=intense/severe) for (1) the number of wheals (hives) and (2) itch intensity over the previous 12 hours, ranges from 0 to 6, and is measured twice daily (morning and evening). The Baseline score is the sum of the daily urticarial activity scores over the 7 days prior to the first treatment. A higher urticarial activity score indicates more urticaria activity.
Time Frame: Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Percentage of participants | 11.3 | 26.0 | 40.0 | 51.9
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 75 mg groups. The p-value was not evaluated for statistical significance in accordance with the type I error rate control plan; Test type: Superiority or Other; p = 0.0148, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)

6. Secondary Outcome: Percentage of Weekly Itch Severity Score MID Responders at Week 12
Description: The percentage of participants with an itch severity score at 12 Weeks at least 5 points lower than at Baseline.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Percentage of participants | 36.3 | 55.8 | 56.3 | 75.3
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0226, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 1, analysis 1]

7. Secondary Outcome: Change From Baseline to Week 12 in the Weekly Size of the Largest Hive Score
Description: The weekly size of the largest hive score is the sum of the daily size of the largest hive scores over 7 days and ranges from 0 to 21. The daily size of the largest hive score is assessed twice daily (morning and evening) on a scale of 0 (none) to 3 (> 2.5 cm). The daily size of the largest hive score is the average of the morning and evening scores. The Baseline weekly size of the largest hive score is calculated over the 7 days prior to the first treatment. A higher score indicates larger hives. A negative change score indicates a reduction in hive size.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Units on a scale | -3.93 (5.44) | -6.20 (6.29) | -6.96 (6.68) | -9.79 (6.66)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.0124, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline weekly size of largest hive score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = -2.34, 95% CI 2-sided [-4.17 to -0.51]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.0012, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = -3.16, 95% CI 2-sided [-5.05 to -1.27]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 7, analysis 1]; Least squares mean difference = -5.73, 95% CI 2-sided [-7.59 to -3.87]

8. Secondary Outcome: Change From Baseline in the Overall Dermatology Life Quality Index (DLQI) Score at Week 12
Description: The DLQI is a 10-item dermatology-specific health-related quality of life measure. Patients rated their dermatology symptoms as well as the impact of their skin condition on various aspects of their lives on a scale of 0 (Not at all) to 3 (Very much). The overall DLQI is the sum of the responses to the 10 items and ranges from 0 to 30. A lower score indicates a better quality of life. A negative change score indicates improvement.
Time Frame: Baseline to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 62 | 66 | 63 | 72
Units on a scale | -6.13 (6.25) | -6.33 (6.08) | -8.00 (7.24) | -10.29 (7.23)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.7956, ANCOVA — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline overall DLQI score (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg); Least squares mean difference = 0.26, 95% CI 2-sided [-1.76 to 2.28]
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups; Test type: Superiority or Other; p = 0.2286, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 8, analysis 1]; Least squares mean difference = -1.31, 95% CI 2-sided [-3.46 to 0.84]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 8, analysis 1]; Least squares mean difference = -4.08, 95% CI 2-sided [-5.96 to -2.20]

9. Secondary Outcome: Percentage of Angioedema-free Days From Week 4 to Week 12
Description: The percentage of angioedema-free days from Weeks 4 to 12 was defined as the number of days for which a patient responded "No" to the angioedema question in the daily diary divided by the total number of days with a non-missing diary entry, starting at the Week 4 visit and ending the day prior to the Week 12 visit.
Time Frame: Week 4 to Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 66 | 69 | 70 | 74
Percentage | 88.2 (19.4) | 86.5 (28.4) | 89.6 (20.6) | 96.1 (11.3)
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4867, Stratified Wilcoxon — [p-value comment as in outcome 2, analysis 1]; Stratification variables included in the analysis were presence of angioedema at baseline (yes vs no) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 150 mg groups. The p-value was not evaluated for statistical significance in accordance with the type I error rate control plan; Test type: Superiority or Other; p = 0.1747, Stratified Wilcoxon — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 9, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Stratified Wilcoxon — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 9, analysis 1]

10. Secondary Outcome: Percentage of Complete Responders (UAS7 = 0) at Week 12
Description: A complete responder was defined as a participant with a UAS7 score = 0 at Week 12.
Time Frame: Week 12
Population: Modified intent-to-treat population: All randomized patients who received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Number analyzed (Participants) | 80 | 77 | 80 | 81
Percentage of participants | 8.8 | 11.7 | 15.0 | 35.8
Statistical Analysis 1: Comparison: Placebo vs Omalizumab 75 mg; [analysis description as in outcome 5, analysis 1]; Test type: Superiority or Other; p = 0.4580, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 2: Comparison: Placebo vs Omalizumab 150 mg; [analysis description as in outcome 9, analysis 2]; Test type: Superiority or Other; p = 0.2087, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)
Statistical Analysis 3: Comparison: Placebo vs Omalizumab 300 mg; The null hypothesis was that there was no difference between the placebo and the omalizumab 300 mg groups; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; Covariates included in the analysis were baseline UAS7 (< median vs ≥ median) and baseline weight (< 80 kg vs ≥ 80 kg)

ADVERSE EVENTS:
Time Frame: Adverse events were reported starting with the first dose of study drug through the end of the study (up to 40 weeks).
Description: Safety population: All randomized participants who received at least 1 dose of study drug.
Arm/Group | Placebo | Omalizumab 75 mg | Omalizumab 150 mg | Omalizumab 300 mg
Serious Adverse Events (participants affected / at risk) | 5/80 | 2/70 | 5/87 | 2/81
Other Adverse Events (participants affected / at risk) | 38/80 | 37/70 | 46/87 | 40/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Omalizumab 75 mg (N=70) | Omalizumab 150 mg (N=87) | Omalizumab 300 mg (N=81)
Angina unstable (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Shock hypoglycaemic (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=80) | Omalizumab 75 mg (N=70) | Omalizumab 150 mg (N=87) | Omalizumab 300 mg (N=81)
Nasopharyngitis (Infections and infestations) | 17 | 5 | 14 | 10
Sinusitis (Infections and infestations) | 5 | 6 | 7 | 5
Upper respiratory tract infection (Infections and infestations) | 3 | 6 | 4 | 4
Bronchitis (Infections and infestations) | 6 | 5 | 2 | 2
Urinary tract infection (Infections and infestations) | 3 | 3 | 7 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 5 | 4
Headache (Nervous system disorders) | 4 | 5 | 12 | 7
Asthma (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 4 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 5 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3 | 0
Idiopathic urticaria (Skin and subcutaneous tissue disorders) | 4 | 10 | 7 | 11
Urticaria (Skin and subcutaneous tissue disorders) | 8 | 8 | 7 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.